CLINICAL TRIAL: NCT00794703
Title: A Multi-center, Randomized, Open Label, Parallel Study to Evaluate and Compare the Efficacy and Safety of Mycamine® vs Itraconazole Oral Solution for Prophylaxis of Fungal Infections in Patients Undergoing a Hematopoietic Stem Cell Transplant
Brief Title: A Study to Compare Efficacy and Safety of Mycamine® and Itraconazole for Preventing Fungal Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCFGCN02-0
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Fungemia; Fungal Infections
Keywords: Antifungal; micafungin; itraconazole
MeSH Terms: conditions — Fungemia; Mycoses | interventions — Micafungin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Micafungin (Experimental)
  Interventions: Drug: micafungin (Mycamine)
- 2. Itraconazole (Active Comparator)
  Interventions: Drug: itraconazole

INTERVENTIONS:
Drug: micafungin (Mycamine) — Intravenous
  Other Names: Mycamine; FK463
  Arms: 1. Micafungin
Drug: itraconazole — oral
  Other Names: Sporanox
  Arms: 2. Itraconazole

SUMMARY:
The objective of this study is to compare the efficacy and safety between Mycamine and Itraconazole oral solution in preventing invasive fungal infections on autologous(malignant blood diseases) or allogeneic hematopoietic stem cell transplant patients

DETAILED DESCRIPTION:
Dosing of Mycamine or Itraconazole will start at the beginning of the transplant conditioning regimen or within 48 hours after the transplant conditioning regimen, and administration time should be no longer than 42 days

ELIGIBILITY:
Inclusion Criteria:

* Patients at risk of systemic fungal infections due to their immunocompromised state due to one of the following:

  * Patient with a hematologic malignancy undergoing an autologous hematopoietic stem cell transplant
  * Any patient undergoing an allogeneic hematopoietic stem cell transplant

Exclusion Criteria:

* Patients with moderate or severe liver disease, as defined by:

  * AST or ALT greater than 5 times upper limit of normal (ULN), OR;
  * Total bilirubin greater than 2.5 times ULN
* Patients with evidence of a deeply invasive or disseminated fungal infection at time of enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Treatment success rate (fungal breakthrough rate) | At the end of the study

SECONDARY OUTCOMES:
Incidence of proven or probable invasive fungal infection | Throughout the study period
The usage rate of systemic antifungal agents | During 4 weeks after the administration
Time to treatment failure | During the study period
Assessment of Adverse events, Laboratory examinations and vital signs evaluation | Throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (10):
- China (10):
  - Fuzhou, Fujian
  - Wuhan, Hubei
  - Chengdu, Sichuan
  - Hangzhou, Zhejiang
  - Beijing
  - Jiangsu
  - Nanning
  - Shanghai
  - Tianjin
  - Xi'an

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang X, Chen H, Han M, Zou P, Wu D, Lai Y, Huang H, Chen X, Liu T, Zhu H, Wang J, Hu J. Multicenter, randomized, open-label study comparing the efficacy and safety of micafungin versus itraconazole for prophylaxis of invasive fungal infections in patients undergoing hematopoietic stem cell transplant. Biol Blood Marrow Transplant. 2012 Oct;18(10):1509-16. doi: 10.1016/j.bbmt.2012.03.014. Epub 2012 Mar 30. PMID 22469884
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=MCFGCN02-0